Study Title: Building Partnerships with First Responders to Explore Strategies

to Improve Delivery and Access of Mental Health Services

NCT Number: NCT03801408

**Principal Investigator:** Sara Jones, PhD, APRN, PMHNP-BC

**Assistant Professor** 

University of Arkansas for Medical Sciences, College of Nursing

4301 W. Markham Street, Slot # 529

Little Rock, AR 72205 Telephone: 501-526-7846 Email: SLJones@uams.edu

**Sub-investigators:** Jean McSweeney, PhD, RN

Professor and Associate Dean for Research, College of Nursing

Telephone: 501-296-1982

Email: McSweeneyJeanC@uams.edu

Geoffrey Curran, PhD,

Professor, Departments of Pharmacy Practice and Psychiatry

Director, Center for Implementation Research

Telephone: 501-686-7610

Email: CurranGeoffreyM@uams.edu

Virginia Austin, MS, LCSW

Research Program Manager, UAMS College of Nursing

Telephone: 501-603-3518 Email: <u>VAAustin@uams.edu</u>

**Study location:** University of Arkansas for Medical Sciences

4301 W. Markham Street, Slot # 529

Little Rock, AR 72205

**Support Funding:** NIH/NIMH

Date: July 20, 2020

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

# **Table of Contents**

Date: July 20, 2020

| Table of Contents |
|----------------------------------------|
| Background and Rationale |
| Specific Aims |
| Study Design and Procedures |
| Study Population |
| Inclusion Criteria |
| Exclusion Criteria |
| Risks and Benefits |
| Data Handling and Recordkeeping |
| Data Analysis |
| Phase 2 |
| Ethical Considerations |
| Implications and Dissemination of Data |
| References |

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

## **Background and Rationale**

Sentinel events, such as the attacks on September 11, 2001 (9/11), have focused attention on the magnitude of traumatic exposure experienced by first responders (FRs). <sup>11</sup> In the United States (U.S.), firefighters and EMT/paramedics respond to more than 50 million emergency calls annually. <sup>1,2</sup> Although many FRs serve entire careers without responding to events like those of 9/11, the daily operations and experiences they expect and accept as part of their jobs expose them to a myriad of traumatic events (e.g. fatal vehicle accidents, suicides, school shootings). The nature, frequency, and intensity of duty-related traumatic exposures place FRs at significant risk for developing mental health (MH) problems. <sup>3</sup>

An estimated 18-37% of FRs worldwide meet criteria for posttraumatic stress disorder (PTSD),<sup>8</sup> a rate similar to that among military veterans (10-31%),<sup>19</sup> and much higher than that in general populations (8.7%).<sup>4,12,13</sup> MH problems among FRs are not limited to PTSD; prevalence rates for other problems are: 7-22% for depression,<sup>14,15</sup> 4-22% for anxiety,<sup>4,16</sup> 34-56% for binge drinking,<sup>17,18</sup> and 58-70% for sleep problems.<sup>14,19</sup> MH problems can emerge in training<sup>14</sup> and continue long after retirement, with approximately 15% of suicides among FRs occurring in retirees.<sup>20,21</sup> In one study (n=1027), 15.5% of FRs reported at least one suicide attempt during their careers,<sup>5</sup> much higher rates than those in general adult populations (1.9-8.7%).<sup>5,8,22</sup>

However, we were able to locate virtually no published research on rates of help-seeking and service utilization among FRs with MH problems. Less than 40% of the general population who experience MH problems seek help,<sup>6</sup> and help-seeking is expected to be even lower among FRs because of the stigma associated with mental illness and the emphasis that FR culture puts

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

on strength and self-reliance.<sup>5,7</sup> According to published personal accounts, MH problems are

viewed as signs of vulnerability; acknowledging them can lead to mistrust and raise questions

about personal safety of others within FR departments.8 There is apprehension about allowing

"outsiders" into the culture, which creates isolation and inhibits help-seeking. Yet, there is

minimal research to corroborate these personal testimonies. We urgently need to understand

FRs' perspectives about accessing and engaging in MH services to guide development of a MH

service model they will be willing to access and use.

Evidence is scarce regarding FRs' barriers to help-seeking. Two recent studies described

both structural and cultural barriers, such as cost and availability of resources, <sup>23</sup> perceived

accessibly of treatment, and concern about stigma.<sup>24</sup> Hom et al. found that firefighters who

experienced suicidal thoughts/behaviors, but did not utilize services reported more concerns

about reputation and embarrassment than those who did use services.<sup>25</sup> The literature on U.S.

military veterans and law enforcement officers (LEOs), similar cultural groups, provides useful

clues.8 For instance, veterans report barriers to accessing MH services to include concerns about

negative consequences of disclosing MH problems, discomfort with help-seeking, and negative

values/ beliefs regarding MH treatment. 26,27 Strategies to reduce stigma and improve MH care

among veterans suggest the importance of non-stigmatizing language related to MH, anonymity,

and peer-to-peer support. 28 LEOs are concerned that help-seeking indicates weakness; they also

fear loss of confidentiality and threats of job loss. <sup>29,30</sup> Although literature on veterans and LEOs

is suggestive, FRs (as defined by this study) are unique in structural and cultural ways that may

influences help-seeking and require tailored approaches to address their MH problems.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

The need for research and resources to address MH problems among FRs is well recognized

by national FR organizations. The National Fallen Firefighters' Foundation (NFFF), Initiative

13: Psychological Support, emphasizes the need for resources to help FRs cope with duty-related

complications, especially regarding emotional and psychological stress. The 2015 National Fire

Service Research Agenda recommends research to identify individuals who are at high risk for

health problems, especially those related to repeated trauma exposures. In particular, the agenda

gives high priority to efforts to "identify, develop, and refine evidence-based tools and

approaches for behavioral health screening, assessment, and intervention" (p.17).<sup>31</sup> NFFF also

highlights the need for a new model of MH screening and interventions that better reflects the

variability in how FRs respond to traumatic incidents. The importance of tools that reflect

variability is supported by a survey conducted by National Volunteer Fire Council (n=849). Over

75% of firefighters indicated greater willingness to utilize a program that was tailored to their

needs compared to a national suicide hotline. 14 This supports the need for research to develop a

tailored MH service model to support early identification and treatment of FRs' MH problems.<sup>31</sup>

Evidence of the effectiveness of MH services commonly available to FRs is lacking. Many

FR departments offer limited MH services, with the two most common being Critical Incident

Stress Debriefing (CISD) and Employee Assistance Programs (EAPs). However, empirical

evidence for these interventions is inconsistent. CISDs are in-house debriefing sessions

implemented within 72 hours after an incident; the limited published research on CISD does not

provide strong evidence for its effectiveness.<sup>32</sup> Previous studies have shown that CISD can

actually increase the risk of PTSD among those that receive debriefing (OR 2.51; 95% CI 1.24 to

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

5.09). 33,34 Qualitative research regarding this topic is limited to one national study (n=423) that

explored firefighters' perceptions about CISD; some FRs reported CISD to be beneficial, others

found it to be intrusive and distressing.<sup>35</sup> Still, CISD continues to be used by FRs nationwide.<sup>35</sup>

EAPs are outside agencies contracted to provide MH services to FR departments. Although they

are widely used, we were unable to find research on FRs' perceptions of EAPs or their

effectiveness in meeting FRs' MH needs.

**Preliminary Studies (PS)** 

PS#1: Funded by a UAMS College of Nursing intramural grant (January, 2017). The PI used

community engagement to establish partnerships with key FR stakeholders across AR to discuss

FRs' MH-related issues, including the: Director of Emergency Medical Services (EMS), AR

Department of Health; Fire and EMS Coordinator, AR Department of Emergency Management;

President of AR Professional Firefighters Association, local EMS directors, and multiple fire

chiefs statewide (see Letters of Support). They expressed concern about the increased prevalence

of MH problems among their FRs, and attributed the increase in number of suicides and early

retirements over the past decade to MH problems. They also reported a lack of help-seeking even

when MH problems were apparent and EAP and/or CISD were available. All community

partners were highly motivated to address MH problems among FRs, but have lacked resources

and expertise to do so. For example, the President of AR Professional Firefighters Association

reported that they have pushed legislation to address MH issues in the fire service for years, but

have been unsuccessful. These partnerships will be critical to the successful conduct of the

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

proposed research as well as future implementation, dissemination, and sustainability of the

resulting MH service model for FRs.

PS#2: Funded by an International Society of Psychiatric Nursing Foundation Research grant

(March 2017). The specific aims for this ongoing PS are to 1) assess the feasibility of using a

community-engaged approach with FRs, 2) characterize the MH profile of Arkansas' FRs, and 3)

explore individual FRs' perceptions of MH problems and use of MH services, including barriers

and facilitators to help-seeking. To achieve Aim 1, the PI collaborated with PS#1 community

partners to refine recruitment methods; these methods will be used in the proposed study

(described below). Recruitment was successful and resulted in ample and continued access to

this population, including presentations at four FR-related state conferences. To achieve Aim 2,

FRs statewide were invited to complete an anonymous online survey that incorporated brief

assessments of various MH problems, <sup>42</sup> as well as questions addressing demographics and

factors that can pose as potential risk/protective factors (e.g., marital status, military service). 10,42

A total of 220 FRs started the survey and 87% completed it. Of completers, 86% were male and

95% were Caucasian; the average length of time as a FR was 16.2 years; 23% reported a

previous MH diagnosis and 25% reported previous MH treatment. The high rates of self-reported

MH problems found were: 26% for PTSD; 28% for moderate to severe anxiety; 14% for major

(moderate-severe to severe) depression; 20% for harmful/ hazardous drinking; and, 34% for

high-risk for suicidal behaviors, highlighting the need for the proposed study.

To achieve Aim 3, we conducted in-depth, ethnographic interviews with individual FRs.

Thirty-two FRs were interviews; of those interviewed, 36% reported a previous MH diagnosis,

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

and 40% reported previous MH treatment. Experience with Aim 3 demonstrates the willingness

of FRs with MH problems to participate in qualitative research. Grounded theory-informed,

qualitative analytic methods (as described below) were used to identify common themes. The

main the themes included: knowledge, barriers and facilitators to help-seeking, effects of the job

and coping with them, non-duty stressors, pros and cons of existing MH services and delivery

methods, and novel delivery approaches.

**Specific Aims** 

Based on preliminary data and current literature, there is crucial need to reduce barriers to

access and promote engagement in MH services to address FRs' MH needs. To develop an

effective MH service model that will be accessed and used by this high-risk group, we must

understand and incorporate FRs' preferences for MH service and delivery methods. We propose

a two-stage exploratory, qualitative study that will use a statewide community-engagement

approach to conceptualize a MH service model that would motivate FRs to be more engaged in

services. In Stage 1, we will conduct qualitative focus groups (and individuals interviews, as

needed; see below) with firefighters and EMTs/ paramedics across Arkansas. In Stage 2, we will

use a product development process grounded in these findings to conceptualize a MH service

model feasible for implementation in real world settings. (Protocol for Stage 2 will be submitted

for IRB approval at a later time.)

Phase 1-Specific Aim 1: Identify FRs' preferences and priorities regarding MH service and

delivery methods, including the feasibility, acceptability, and value of each method. (Method:

*Qualitative interviews- focus groups and individual)* 

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

Phase 2, Specific Aim 2: Conceptualize a MH service model, in partnership with FRs statewide,

that is applicable, acceptable, and feasible for implementation. (Method: Virtual Delphi group of

consensus formation)

Through this multi-phase work, we will generate the scientific foundation to develop a

comprehensive, MH service model that diverse FRs will be willing to access and use. Based on

FRs preferences and priorities, we expect this model will encompass a range of services, such as

education and awareness initiatives, prevention and screening strategies, and crisis and

maintenance interventions, to meet their MH needs throughout the course of illness.

**Study Design and Procedures** 

This qualitative study will use a statewide community-engagement approach to explore FRs

preferences for MH service and delivery methods. In a community-engagement approach,

researchers form collaborative partnerships with key stakeholders; together, they identify areas

of interest and concern.<sup>45</sup>

Phase 1-Specific Aim 1: Identify FRs' preferences and priorities regarding MH service and

delivery methods, including the feasibility, acceptability, and value of each method.

**Instruments and Measures** 

Prior to starting the focus group/interview, the PI or research associate (RA) will distribute a

one-page document to reference during the informed consent process; the document will describe

the study purpose, procedures, risks, and benefits (Human Subjects Protection); time will be

allowed for questions. Participants will be advised that participating implies consent and they

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

may withdraw at any time. (We received a waiver of documentation of consent for the interviews in PS#2; we will seek the same for this study). Rules of confidentiality will also be discussed.

Following the consent process, participants will be asked to complete a brief form to collect data about demographics (i.e., age group, race/ethnicity, gender) and potential risk/protective factors (e.g., time in service, military service, medical problems).

The PI and/or RA will facilitate the focus group (FG) discussions using a semi-structured question guide (Table 2), which will have undergone review by our community partners. (In addition to content, we will ask them for feedback regarding language, ensuring it is non-stigmatizing.)

To start the group discussion, the PI/RA will use a PowerPoint presentation to highlight the various MH services discussed in the PS interviews. Group participants will be asked to discuss the pros and cons of existing MH services and delivery methods, and novel approaches that

emerged during the interviews. They will be asked to discuss their own experiences related to each; based on their experiences, they will be asked to make recommendations for services/delivery methods that would motivate FRs to be more engaged in services. We will ask them "where to start" when implementing a MH service model; follow-up questions will include probes related to

| Main Question | Which of these services and methods of delivery do you recommend? |
|---|---|
| Probe<br>Questions | What do you like and not like about each of these services and delivery methods? |
| | Do you foresee any additional barrier to using these services? Barriers to implementing them? |
| | Could they be modified/adapted to better fit the first responder culture and environment? |
| | Would you suggest any additional services or methods that we haven't discussed yet? |
| | What do you think we should start with first? |

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

acceptability and feasibility. (Similar methods were effectively used in a study conducted by Co-

investigator Curran and colleagues).<sup>51</sup>

In concluding the FGs, we will offer optional telephone follow-ups to participants who may

be reluctant to express their views in the group. Participants will also receive a blank piece of

paper, along with a web link to an anonymous form in Survey Monkey. Here, they can add

information they may not be comfortable discussing in the FG; text data from these options will

be included in data analysis. Additionally, the PI/RA will record field notes during each FG,

noting information about context, nonverbal communication, and interactions observed during

the FG.<sup>52</sup>

Research Team

The PI is psychiatric advanced practice registered nurse whose qualifications to serve as PI

on this project stem from: 1) well-established community partnerships with FRs across the state;

2) having completed a systematic review and pilot studies related to the MH of FRs<sup>36, 37</sup>; 3)

previous clinical and research experience with individuals that have experienced trauma; and, 4)

interdisciplinary collaboration with experts in the fields of emergency medical services and

qualitative research. Co-I McSweeney is an expert in qualitative methods. She will attend

monthly team meetings to evaluate the FG processes, including development of the FG question

guide and assist in qualitative data analysis (as described in Data Management and Analysis

section). Co-I Curran is an expert in implementation science and has conducted multiple

qualitative studies related to help-seeking and use of MH services. He will attend monthly team

meetings regarding these aspects of study implementation, including the FG method (which was

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

successfully used in his previous studies). The RA is a licensed social worker (LCSW) with over

10 years' experience, and a local volunteer firefighter.

**Study Population** 

Participants will include a convenience sample of firefighters and EMTs/paramedics from

across Arkansas.

Inclusion criteria

• ages 18 and over;

• volunteer and career personnel;

• active, inactive, and retired

Exclusion criteria

• Non-english speaking (due to the nature of FG/interview discussions).

Recruitment

We will use opt-in methods, facilitated by our community partners, to recruit participants.

The PI will visit recruitment sites, provide refreshments, distribute promotional materials, and

discuss long-term study goals. She will send emails to community partners that include study

information, invitations to participate, and suggested text for

email reminders.<sup>50</sup> Partners will then distribute the emails

throughout their departments; the State EMS Director will

distribute through the state EMS registry, which includes all

certified EMT/paramedics in the state. Emails and promotional



Figure 2: Arkansas: Regional Map

Access of Mental Health Services

information will be requested online.

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

materials will instruct FRs to contact the PI or research assistant (RA) by telephone for more study information. They will also have the option to follow a web link (available as a Quick Response [QR] code) where they can read more about the study and/or submit their name (first name, last initial), phone number and/or email address to be contacted with more study information. They will also be asked which region of the state they respond in; no additional

Many community partners are involved in FR-related organizations; she may be invited to present and recruit at state meetings. Some of the departments also distribute monthly/ quarterly newsletters; study information will be published therein (with approval from the administration). The flyer will also be placed on social media sites, such as Facebook and Instagram.

Sampling and Sample Size. An essential part of grounded theory-informed methods is the use of theoretical sampling. <sup>49</sup> In grounded theory research, we do not know the important themes in advance; instead, they emerge and are refined over time as data are collected and analyzed. In general, exploration of a certain theme is stopped when "saturation" is reached, that is, no new themes emerge from the data (discussed below). Therefore, theoretical sampling does not provide a detailed sampling schema or calculation for number of participants beforehand. For this study, we will recruit FRs to participate in up to 25 FGs that will include 5-12 participants per group. Eighteen of these groups will be open to all FRs from different regions across the state. Evidence suggests that call volume and career vs. volunteer service influence FRs' MH. <sup>42</sup>
The 2 most populous regions in Arkansas (Central and Northwest) have higher EMS call volumes and a greater number of career fire/ambulance services than the other 4 regions; the

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

latter are more rural and are served primarily by volunteer fire/ambulance services (Figure 2).

Therefore, we propose to conduct 1) five FGs in each of the two most populous regions

(total=10), and 2) two FGs in each of the other four regions (total=8).

Since the majority of FRs are white males, 1,62 female and minority FRs may be reluctant to

openly discuss MH-related issues in a diverse group. We will conduct a minimum of 2 of the 25

FGs with an ethnically diverse group of females only, and an additional 2 FGs with minorities

only (males and females) (total=4). This will ensure that at least 10-15% of participants are

females and minorities. We will make every effort to recruit these participants from across AR,

but due to the distribution of FRs across AR, we expect these FGs will take place in Central and

Northwest AR.

Sample Size

An essential part of qualitative methods is the use of theoretical sampling. Theoretical

sampling does not provide a detailed sampling schema or calculation for number of participants

beforehand. Instead, exploration of a certain theme is stopped when "saturation" is reached, that

is, no new themes emerge from the data (see Analysis section).

Compensation

Participants will receive a \$25 Walmart gift card upon completion of the FG or interview.

Limitations

A possible barrier to this study may be recruitment concerns. To date, all chiefs contacted

have understood the significance of this study and have agreed to encourage participation.

However, individuals may also be reluctant to participate. During recruitment, we will explain

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

the confidential manner of this study to all potential participants: that is, all data will be

unidentifiable and individual responses will not be shared with employers and administrators.

**Risks and Benefits** 

Adult Minimal Risk: Any activity where the probability and magnitude of harm or discomfort

anticipated in the research is not greater in and of themselves than those ordinarily encountered

in daily life or during the performance of routine physical or psychological examinations or tests.

Participants may experience distress at the time of, or because of the focus group/interview

discussions. Prior to starting participation, they will be advised that if this occurs, they can

choose to stop meet with the PI/RA individually. They will also be advised that the PI/RA may

ask them to discontinue participation or ask to meet afterwards if a significant level of distress is

observed. In meeting with the participant individually, the PI, an experienced psychiatric-mental

health nurse practitioner, or RA, a licensed social worker (LCSW) with over 10 years'

experience, will briefly evaluate him/her and conduct a suicide risk assessment if indicated.

Based on the evaluation, the participant may be referred for services, including (but not limited

to) a local emergency department (if currently experiencing active suicidal ideations), the locally

contracted EAP, or other MH services.

The PI has received permission from various MH providers, including therapists and nurse

practitioners, which have agreed to be listed as an available resource for the purposes of this

study. This list of compiled resources, along with a list of phone numbers, will be available at all

sites and online at the link provided on the flyer. The phone numbers will include 911 (for

emergencies), local and/or national suicide hotline numbers, and the PI's phone number. If

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

called, the PI (or consulting provider) will conduct an appropriate evaluation, including a suicide

assessment, and make referrals as appropriate (as mentioned above). Documentation and follow-

up will also be completed as applicable. This information (available resources and phone

numbers) will also be provided upon completion of the group/interview and maintained online at

the link provided in the email.

Suicide Risk Assessment and referral. The PI/RA will use the Suicide Assessment Five-step

Evaluation and Triage (SAFE-T) for Mental Health Professionals to assess risk of suicide and

make referrals (uploaded in attachments). SAFE-T is a resource recommended by SAMSHA and

published by the National Suicide Prevention Lifeline. This 5-step assessment guides the

provider to: 1) identify risk factors, 2) identify protective factors, 3) conduct suicide inquiry, 4)

determine risk level/intervention, and 5) document.

To reduce risk of breach of confidentiality, audio-recordings of the focus groups/interviews

will be stored in a locked filing cabinet and all transcriptions will be electronically documented.

All electronic data will be maintained on a password-protected server to which only the research

team will have access. The HIPAA compliant version of SurveyMonkey will be purchased; only

aggregate data from the surveys will be reported.

Benefits

There may be no personal benefits to the individual participants at the time of the study. It is

possible, however, that participating in this study will increase participants' awareness of, and

decrease stigma related to, mental and substance use disorders, which may prompt some to seek

services. Further, findings from this study will guide future studies to develop tailored prevention

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

and treatment strategies that are accessible across Arkansas to improve the overall mental and

emotional well-being of FRs.

**Data Handling and Recordkeeping** 

The PI will carefully monitor study procedures to protect the safety of research subjects, the

quality of the data and the integrity of the study. All data will be recorded without identifiers and

will be anonymous. Audio-recordings will be stored in a locked filing cabinet and all

transcriptions will be electronically documented. All electronic data will be maintained o on a

password-protected UAMS server, both located behind locked doors in a restricted access area of

the UAMS campus. Only the PI, Co-Is, and Research Assistant (to be determined) will have

access to the data.

**Data Analysis** 

The RA will enter quantitative participant data (i.e. demographics, risk/protective factors)

into SPSS (V24).53 Data will be analyzed using standard statistical techniques to summarize data

distributions and to model associations among risk and status variables. FGs and interviews will

be audio recorded, transcribed verbatim, and entered into a professional software program

designed to facilitate the data analysis process and produce an audit trail.<sup>54</sup> Data submitted online

will also be entered.

We will analyze data using grounded theory-informed methods of content analysis and

constant comparison. 43 Content analysis is a systematic, objective analysis designed to identify

key words, phrases, and topics, which guides top-level coding.<sup>55</sup> This process is followed by

constant comparison, second-level coding, an iterative process designed to identify common

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

themes by comparing one set of data to another. <sup>49</sup> We will also use this process to compare data across sub-groups (e.g. urban/rural, male/female). The PI has experience in qualitative methods;

both co-Is have expertise in qualitative methods; and the RA will be trained in these methods.

Top-level coding. The PI, co-I (McSweeney), and RA will independently review the transcripts from the first 3 FGs. Using content analysis, similar data from these transcripts will be identified, grouped, and assigned a label, referred to as a code. 47 These codes will reflect the themes and subject areas that, by virtue of their recurrent nature, seem most important to answering the key research questions. The research team will meet to compare coding and reach consensus on coding that differs. This process will continue with additional transcripts until they reach consensus on a set of initial top-level codes and definitions for each code, which will comprise the *code book*. This process will ensure inter-rater reliability, that is, consistency in coding.<sup>56</sup> Thereafter, the PI and RA will individually code the remaining transcripts using the codebook. To ensure coding consistency, they will review each other's work monthly and meet to discuss and resolve any differences. In the event that new themes emerge after the codebook is

Second-level coding. Second-level coding is a process to further refine the constructs indicated by top-level codes. The final codebook will be used to "sub-code" data within each code. That is, data within codes will be compared across transcripts to find similarities, differences, associations, and relationships to determine patterns and thematic categories,

agreed upon, the research team will meet again to define emerging codes; previously coded

transcripts will be recoded to reflect the additions(s).

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

creating these sub-themes. The process of inter-rater reliability (discussed above) will be used to

establish reliability.

Saturation. In general, exploration of a certain theme is stopped when "saturation" is

reached, that is, when no new concepts or properties emerge from the data after the thematic

categories are identified. Given the potential size of the overall sample from the FGs (n=132-

220) and individual interviews (n=44), we will have no difficulty in achieving overall saturation.

Additionally, based on the anticipated diversity of the FGs, we expect to be able to achieve

saturation for both urban (n=60-100) and rural (n=48-80) FRs, as well as for female (n=12-20)

and minority (n=12-20) FRs. We will use standard qualitative guidelines for trustworthiness by

Lincoln and Guba (1985) to maximize the project's validity and reliability.<sup>57</sup> A data table will be

constructed to provide an audit trail that identifies the thematic categories, frequencies of

explanations, and examples of raw data that exemplify each theme. The field notes recorded by

the RA will also be used in this iterative analysis process.

Phase 2, Specific Aim 2: Conceptualize a MH service model, in partnership with FRs

statewide, that is applicable, acceptable, and feasible for implementation.

Product development activity: Delphi technique

After all focus groups have been analyzed, we will initiate a series of product development

activities. We will use a virtual Delphi technique of consensus formation to conceptualize a MH

service model that is acceptable to FRs and feasible to implement in real world settings. This

method has been successful in fostering a sense of ownership and the engagement of diverse

stakeholders in an iterative decision-making process.<sup>58</sup>

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

### **Participants**

We will invite individuals from our community partners (i.e., Arkansas Department of Health, Professional Firefighters Association, etc.) to participate in these Delphi groups, as well as a minimum of 12 diverse FRs who participated in the Phase 1 focus groups. We will aim to include participants from all 6 regions across the state (see page 12). In this way, we will capture the perspectives of both administrative and in-line FRs.

#### **Procedures**

Due to extended proximities and current COVID related guidelines, all discussions will be conducted virtually using Zoom. The initial meeting with be conducted by the PI and RA. The PI will explain the discussion panel's purpose and procedures, including the process, timeline, and expectations. Then, the RA will distribute a handout that briefly describes existing MH services and delivery methods; she will review the Aim 1 findings, including the recommendations and priorities that arose from the groups. After the first meeting, the PI and RA will compile results of the discussion to conceptualize a MH education program. Then, this information will be disseminated to the FR panel for review prior to the next meeting. To allow all individuals to privately agree or disagree with each, a survey will be distributed via Survey Monkey that includes the essential components discussed in the group. Each individual will indicate if they agree or disagree and be able to write additional comments if needed.

The subsequent meetings will aim at reaching consensus on all components of the program.

The RA will lead a series of discussions every other week via Zoom, covering the essential components of a MH service model, including (but not limited to) implementation and

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

engagement strategies, feasibility, and outcome measures. They will also discuss how to meet the

diverse needs within FR populations if differences emerge (e.g. fire vs. ambulance services;

urban vs. rural communities) so that the service model will be generalizable to all FRs.

Following each meeting, we will aim for consensus on the key components discussed during the

group using the survey method discussed above. This technique will allow us to confirm and

document that we have reached consensus.

When employing a Delphi technique, each round of discussion will involve up to three

iterations of deliberations that will seek agreement on essential components of a MH service

model. We will plan to have a minimum of 5 meetings: one for introduction, three for discussion

and deliberations, and one for final presentation. Using multiple rounds of deliberation, along

with a pre-set percentage of agreement, will facilitate a stable and reliable consensus-building

process. In the remote chance that consensus is not reached, we will schedule an additional

called meeting to additional to further discuss and deliberate

We estimate to have a total of 22-24 participants in the Delphi activities. Upon inviting

participants, we will ask them to agree only if they can commit to all meetings, with an

allowance of 1 absence, to assure quorum. Specifically, we will use a minimal consensus level of

75% panel agreement for each component.<sup>60</sup>

Compensation

First responders and associated agencies are already strained with the current pandemic, so

we want to adequately compensate them for their time. Those that commit to and attend at least

4/5 meetings will receive a \$50 Walmart gift card.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

**Ethical Considerations** 

This study will be conducted in accordance with all applicable government regulations and

University of Arkansas for Medical Sciences research policies and procedures. This protocol and

any amendments will be submitted and approved by the UAMS Institutional Review Board

(IRB) to conduct the study. The PI will carefully monitor study procedures to protect the safety

of participants, the quality of the data, and the integrity of the study.

A waiver of documentation of consent is also requested. We will use an IRB-approved

study information sheet to discuss the study and complete the consent process before beginning

the focus groups and interviews. All participants will be provided with an information sheet that

describes this study and provides sufficient information in language suitable for them to make an

informed decision about their participation in this study. The researcher will thoroughly explain

each element of the document and outline the risks and benefits, and requirements of the study.

Questions regarding participation will be answered, no coercion or undue influence will be used,

and participants can leave the group or stop the interview at any time. The informed consent

process will be documented in a process note for each group/interview.

If at any time there is concern that child or elder abuse has possibly occurred, or a participant

discloses a desire to harm self or others, it will be reported to the appropriate authorities.

Implications and Dissemination of Data

Based on information generated by this project, we will pursue a multi-stage research

agenda. Using this study's findings, the next step will be to develop a tailored MH service model

consisting of services and delivery methods that can be generalizable to FRs statewide, and to

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

pilot test it for feasibility and acceptability. To do so, we will apply for funding, such as an R34 through the NIMH Division of Services and Intervention Research. Future research will include a full-scale trial of the model statewide, revised based on pilot results, and then a hybrid effectiveness-implementation trial.

Results of this study may be used for presentations, posters, or publications. The publications will not contain any identifiable information that could be linked to a participant. Dissemination of findings to FRs and MH providers through publications and conferences can extend to national arenas to better meet the needs of all FRs. With continued efforts and partnerships, findings can be integrated into policy and funding-related decisions to sustain the delivery of high-quality MH services for FRs in Arkansas and across the nation.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

#### References

- 1. Hinds-Aldrich M, Knight M, Nicolosi A, Evarts B. *National fire data survey: Findings on the state of the existing american fire data ecosystem*. Quincy, MA: National Fire Protection Association; 2017.
- McCallion T. NASEMSO Survey provides snapshot of EMS Industry. J Emerg Med Servs. November, 2011.
- 3. Haugen PT, Evces M, Weiss DS. Treating posttraumatic stress disorder in first responders: A systematic review. *Clin Psych Rev.* 2012; 32(5):370-380.
- 4. Meyer EC, Zimering R, Daly E, Knight J, Kamholz BW, Gulliver SB. Predictors of posttraumatic stress disorder and other psychological symptoms in trauma-exposed firefighters. *Psychol Serv.* 2012;9(1):1-15.
- 5. Erich J. Earlier than too late: Stopping stress and suicide among emergency personnel. *EMS World*. November, 2014.
- 6. Institute of Medicine. *Psychosocial interventions for mental and substance use disorders: A framework for establishing evidence-based standards*. National Academy of Sciences; 2015.
- 7. National Volunteer Fire Council (NVFC). Suicide in the fire and emergency services:

  Adopting a proactive approach to behavioral health awareness and suicide prevention.

  Greenbelt, MD: NVFC; 2008.
- 8. Henderson SN, Van Hasselt VB, LeDuc TJ, Couwels J. Firefighter suicide: Understanding cultural challenges for mental health professionals. *Prof Psych: Research and Practice*. 2016;47(3):224-230.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

9. Wilmoth J. Trouble in mind. National Fire Protection Association Journal. May, 2014.

- 10. Pescosolido BA, Gardner CB, Lubell KM. How people get into mental health services: Stories of choice, coercion and "muddling through" from "first-timers." Soc Sci Med. 1998;46(2):275-286.
- 11. Benedek DM, Fullerton C, Ursano RJ. First responders: Mental health consequences of natural and human-made disasters for public health and public safety workers. *Annu Rev Publ Health*. 2007;28:55-68.
- 12. American Psychiatric Association (APA). *Diagnostic and Statistical Manual of Mental Disorders (DSM-5)*. 5 ed. Washington, DC: American Psychiatric Publishing; 2013.
- 13. National Institutes of Health (NIH). PTSD: Growing Epidemic. *NIH Medline Plus*. 2009;4(1):10-14.
- 14. Carey MG, Al-Zaiti SS, Dean GE, Sessanna L, Finnell DS. Sleep problems, depression, substance use, social bonding, and quality of life in professional firefighters. *J Occup Environ Med.* 2011;53(8):928-933.
- 15. Fullerton CS, Ursano RJ, Wang L. Acute stress disorder, posttraumatic stress disorder, and depression in disaster or rescue workers. *Am J Psychiatry*. 2004;161(8):1370-1376.
- 16. Bennett P, Williams Y, Page N, Hood K, Woollard M. Levels of mental health problems among UK emergency ambulance workers. *Emerg Med J.* 2004;21(2):235-236.
- 17. Piazza-Gardner AK, Barry AE, Chaney E, Dodd V, Weiler R, Delisle A. Covariates of alcohol consumption among career firefighters. *Occup Med (Lond)*. 2014;64(8):580-582.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

18. Haddock CK, Day RS, Poston WS, Jahnke SA, Jitnarin N. Alcohol use and caloric intake from alcohol in a national cohort of U.S. career firefighters. *J Stud Alcohol Drugs*. 2015;76(3):360-366.

- 19. Courtney JA, Francis AJ, Paxton SJ. Caring for the country: fatigue, sleep and mental health in Australian rural paramedic shiftworkers. *J Community Health*. 2013;38(1):178-186.
- 20. Fjeldheim CB, Nothling J, Pretorius K, et al. Trauma exposure, posttraumatic stress disorder and the effect of explanatory variables in paramedic trainees. *BMC Emerg Med.* 2014;14:11.
- 21. Firefighters Behavioral Heatlh Alliance. http://www.ffbha.org/what-are-these-numbers/.
  Accessed June 6, 2017.
- 22. Stanley IH, Hom MA, Hagan CR, Joiner TE. Career prevalence and correlates of suicidal thoughts and behaviors among firefighters. *J Affect Disorders*. 2015;187:163-171.
- 23. Stanley IH, Boffa JW, Hom MA, Kimbrel NA, Joiner TE. Differences in psychiatric symptoms and barriers to mental health care between volunteer and career firefighters. *Psychiatry Res.* 2017;247:236-42.
- 24. Kim JE, Dager SR, Jeong HS, et al. Firefighters, posttraumatic stress disorder, and barriers to treatment: Results from a nationwide total population survey. *PLoS One* 2018;13(1):e0190630.
- 25. Hom MA, Stanley IH, Ringer FB, Joiner TE. Mental Health Service Use Among Firefighters With Suicidal Thoughts and Behaviors. *Psychiatr Serv* 2016;67(6):688-91.
- 26. Ouimette P, Vogt D, Wade M, et al. Perceived barriers to care among veterans health administration patients with posttraumatic stress disorder. *Psychol Serv.* 2011;8(3):212-23.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

27. Valenstein M, Gorman L, Blow AJ, et al. Reported barriers to mental health care in three samples of U.S. Army National Guard soldiers at three time points. *J Traum Stress*. 2014;27(4):406-414.

- 28. Schreiber M, McEnany GP. Stigma, American military personnel and mental health care: Challenges from Iraq and Afghanistan. *J Mental Health* 2015;24(1):54-59.
- 29. Dowling FG, Moynihan G, Genet B, Lewis J. A peer-based assistance program for officers with the New York City Police Department: report of the effects of Sept. 11, 2001. *Am J Psychiatry* 2006;163(1):151-153.
- 30. Miller L. Practical Police Psychology. Springfield, IL: Charles C. Thomas, Publisher; 2006.
- 31. National Fallen Firefighters Foundation. *Everyone Goes Home: 16 firefighter life safety initiatives*. https://www.everyonegoeshome.com/16-initiatives/. Accessed March 7, 2018.
- 32. Harris MB, Balo-flu M, Stacks JR. Mental health of trauma-exposed firefighters and critical incident stress debriefing. *J Loss Trauma*. 2002;7(3):223-238.
- 33. van Emmerik AA, Kamphuis JH, Hulsbosch AM, Emmelkamp PM. Single session debriefing after psychological trauma: A meta-analysis. *Lancet*. 2002;360(9335):766-71.
- 34. Rose S, Bisson J, Churchill R, Wessely S. Psychological debriefing for preventing post traumatic stress disorder (PTSD). *Cochrane Database Syst Rev.* 2002;(2):CD000560.
- 35. Jahnke SA, Gist R, Poston WS, Haddock CK. Behavioral health interventions in the fire service: Stories from the firehouse. *J Workplace Beh Health*. 2014;29(2):113-126.
- 36. Jones, S. Describing the mental health profile of first responders: A systematic review. *J Amer Psych Nur Assoc.* 2017; 23(3), 200-214. doi: 10.1177/1078390317695266

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

37. Jones S, Nagel C, McSweeney J, Curran G. Prevalence and correlates of psychiatric symptoms among first responders in a rural state. *Arch of Psych Nurs*. 2018. doi: 10.1016/j.apnu.2018.06.007

- 38. Penn, CL. Arkansas trauma system & related measures saving lives, improving stats. *J Ar Med Soc.* 2016;112(11):198-201.
- 39. U.S.Department of Health and Human Services, Health Resources & Services

  Administration. *Health professional shortage areas and medically underserved*areas/populations. https://datawarehouse.hrsa.gov/tools/analyzers/ MuaSearchResults.aspx.

  Accessed March 8, 2018.
- 40. United Health Foundation. *America's health rankings*. www.americashealthrankings.org/ Accessed March 8, 2018.
- 41. Center for Disease Control (CDC). *Mortality in the United States: 2015*. www.cdc.gov/nchs/products/nvsr.htm. Accessed March 8, 2018.
- 42. Jones S. Describing the mental health profile of first responders: A systematic review. *J Am Psych Nurses*. 2017;23(3):200-14.
- 43. Silber H, Litteljohn A, Leibold J. Comparing different types of web surveys: Examining drop-outs, non-resonse and social desirability. *Metodoloski zvezki- Advnaces in Methology and Statistics*. 2013;10(2):121-143.
- 44. FluidSurveys Team. Response rate statistics for online surveys- What numbers should you be aiming for? http://fluidsurveys.com/university/response-rate-statistics-online-surveys-aiming/. Accessed March 8, 2018.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

45. Fawcett SB, Paine-Andrews A, Francisco VT, et al. Using empowerment theory in collaborative partnerships for community health and development. *Am J Community Psychol*. 1995;23(5):677-697.

- 46. National Institute of Mental Health. *NIMH Strategic Plan for Research: Highlight: What Is A Target*? https://www.nimh.nih.gov/about/strategic-planning-reports/highlights/highlight-what-is-a-target.shtml. Accessed March 7, 2018.
- 47. Krueger RA. Focus groups: A practical guide for applied research. (2 ed.). Thousand Oaks, CA: Sage Publications; 1994.
- 48. Streubert H, Carpenter D. *Qualitative research in nursing: Advancing the humanistic imperative*. (2 ed.). Philadelphia, PA: Lippincott; 1999.
- 49. Glaser BG, Strauss AL. *The discovery of grounded gheory: Strategies for qualitative research*. Chicago, IL: Aldine Publishing; 1967.
- 50. Deutskens E, De Ruyer K, Wetzels M, Oosterveld P. Response rate and response quality of internet-based surveys: An experimental study. *Marketing Letter*. 2004;15(1):21-36.
- 51. Medley J, Cheney AMAT, Grubbs K, et al. The Impact of the Psychological Sequela of Trauma on Veterans Seeking Higher Education. *J Postsecond Educ Disabil*. 2017;30(1):83-96.
- 52. Munhall P. *Nursing Research: A Qualitative Perspective*. 4 ed. Sudbury, MA: Jones and Bartlett Publishers; 2007.
- 53. International Business Machines Corporation (IBM). Statistical Package for the Social Sciences (SPSS). 2015.

Access of Mental Health Services

PI: Sara Jones, PhD, APRN

Institution: University of Arkansas for Medical Sciences

Sponsor: NIH/NIMH

55. Morse JM, Field PA. *Qualitative research methods for health professionals*. (2 ed.). London: Sage; 1995.

- 56. Symon G, Castro CA. *Qualitative methods and analysis in organizational research: A practical guide*. London: SAGE Publications; 1998.
- 57. Lincoln YS, Guba EG. Naturalistic inquiry. Beverly Hills, CA: Sage; 1985.
- 58. Rideout C, Gil R, Browne R, et al. Using the Delphi and snow card techniques to build consensus among diverse community and academic stakeholders. *Prog Community Health Partnersh.* 2013;7(3):331-339.
- 59. Asselin M, Harper M. Revisiting the Delphi technique: Implications for nursing professional development. *J Nurses Prof Dev.* 2014;30(1):11-15.
- 60. Keeney S, Hasson F, McKenna H. Consulting the oracle: Ten lessons from using the Delphi technique in nursing research. *J Adv Nurs*. 2006;53(2):205-212.
- 61. United States Census Bureau. *QuickFacts: Arkansas (July 2015)*. https://www.census.gov/quickfacts/table/ PST045216/00. Accessed March 8, 2018.
- 62. National Highway Traffic Safety Administration. EMS Workforce for the 21st Centeruy: A National Assessment (June 2008).

https://www.ems.gov/pdf/EMSWorkforceReport\_June2008.pdf. Accessed March 8, 2018.